CLINICAL TRIAL: NCT00006177
Title: The Phenomenology and Neurophysiology of Affective Dysregulation in Children and Adolescents With Bipolar Disorder
Brief Title: Child & Adolescent Bipolar Disorder Brain Imaging and Treatment Study
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000198; 00-M-0198
Record Dates: First submitted 2000-08-12; First posted 2000-08-14 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03-08

CONDITIONS: Bipolar Disorder; Mood Disorders; Attention Deficit Hyerpactivity Disorder
Keywords: Emotion; Affective Neuroscience; Bipolar Disorder; Child; Child Bipolar; Natural History; BPD; Adolescent Bipolar
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Adult bipolar patients: Adult bipolar patients
- Adult Extended Relatives of BD probands: Adult Extended Relatives of BD probands
- Bipolar Children and Youth: Bipolar Children and Youth
- Child/Adolescent Extended Relatives of BD probands: Child/Adolescent Extended Relatives of BD probands
- Children with ADHD only (controls): Children with ADHD only (controls)
- First degree relatives of BD patients: First degree relatives of BD patients
- Healthy volunteer adults (parents or not): Healthy volunteer adults (parents or not)
- Healthy volunteer children and youth: Healthy volunteer children and youth

SUMMARY:
This research protocol seeks to learn more about bipolar disorder in children and adolescents ages 6-17. Researchers will describe the moods and behaviors of children with bipolar disorder and use specialized testing and brain imaging to learn about specific brain changes associated with the disorder. This protocol studies children who have been diagnosed with bipolar disorder, and those who have a sibling or parent with bipolar disorder and are thus considered "at risk" for developing the disorder.

DETAILED DESCRIPTION:
Objective:

For this protocol we define Bipolar Spectrum disorders (BSD) as the propensity to have a manic episode by having Bipolar Disorder or Substance/Medication-Induced Bipolar and Related Disorder. BSD in children and adolescents is receiving increased research attention, but important questions remain about its developmental trajectory, phenomenology and behavioral correlates, and little is known about its underlying neural mechanisms. In its study of youth with BSD, this study has three objectives:

1. to use longitudinal techniques to characterize the clinical and physiological manifestations of pediatric BSD, and to use cross-sectional techniques (e.g., comparing children and adults with BSD on these measures) to provide preliminary data to guide such longitudinal studies
2. to identify and follow longitudinally behavioral, neuropsychological, neurophysiological, and neuroanatomical correlates of pediatric BSD, and compare to children with chronic irritability and hyperarousal symptoms (severe mood dysregulation, SMD, as outlined in protocol 02-M-0021), youth with attention deficit hyperactivity disorder (ADHD), and typically developing youth.
3. to examine genetic and familial correlates of pediatric BSD

Study population:

There are 11 separate populations being studied in this protocol:

1. Children and adolescents between the ages of 6-17 years old who meet criteria for BSD.
2. Adults between the ages of 18-58 years old who meet criteria for BD, including those age 18-25 with BSD.
3. Control populations of: a) Healthy volunteer children and adolescents between the ages of 3-17 years old, b) Parents of healthy volunteer children or healthy adults in research, c) Children 8-17 years old with attention deficit hyperactivity disorder (ADHD), who do not have a mood disorder.
4. First and second-degree biological relatives of those in (B.1) or (B.2), above, and are between 3-58 years old.
5. A subgroup of these cohorts will be Old Order Amish individuals who fulfill eligibility for (1), (2), (3a), (3b), or (4).

Design:

For children and adolescents with BSD (i.e. Bipolar Disorder or those with Substance/Medication-Induced Bipolar and Related Disorder), this study is an outpatient characterization and longitudinal follow-along design. Once determined to be eligible, individuals come for an initial assessment, and then at varying intervals they return for clinical interviews, behavioral tasks, and structural and functional MRI.

For children and adolescents who are relatives of individuals with BSD, this is an outpatient follow-along design during which individuals come for an outpatient assessment and at 2-year intervals for clinical interviews, behavioral tasks, and structural and functional MRI.

For healthy volunteer children, children with only ADHD, adults with BD, and parents of healthy volunteer children, this study is an outpatient cross-sectional study that includes clinical interviews, behavioral tasks, and structural and functional MRI.

For all others, individuals come to NIH for clinical interviews, behavioral tasks, and MRI.

For most individuals in the Amish community, the investigation occurs in the field, where they receive clinical interviews and behavioral tasks. Some may choose to come to the NIH to participate in behavioral testing and MRI.

For all individuals, genetic material from saliva or blood is obtained under protocol 01-M-0254.

Outcome measures:

This study will examine between group differences in clinical, behavioral, genetic, neuroanatomical, and neurophysiological variables in individuals with BSD, their relatives, and healthy volunteers. Findings in children with BSD will also be compared to those with severe mood dysregulation, sometimes called a broad phenotype of pediatric BD, recruited under protocol 02-M-0021 (Nottelman, 2001).

Longitudinal clinical, behavioral, and neuroanatomical data will also be obtained.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Inclusion and exclusion criteria for each group are outlined below. The total accrual ceiling is 2050, including subjects of both sexes, made up of the following 11 populations:

Pediatric patients with bipolar disorder or SMIBRD:

INCLUSION CRITERIA:

* Age 6-17
* Meet DSM criteria for BD
* Have a primary caregiver who can accompany him or her on trips to NIMH and provide reliable history and information.
* Have a psychiatrist who provides clinical care for their BSD.
* Be able to complete self-rating forms and to cooperate with other study procedures.

EXCLUSION CRITERIA:

* I.Q. < 70
* Autistic disorder or more than mild autism spectrum disorder;
* Psychosis that interferes with the child s capacity to understand and comply with study procedures
* Unstable medical illness (e.g. severe asthma)
* Medical illness that could cause the symptoms of BSD (e.g. multiple sclerosis, thyroid disease)
* Pregnancy
* Substance abuse within two months of the initial evaluation, since alcohol and abused substances interfere with interpretation of fMRI and cognitive task data.
* NIMH IRP Employee family member

Adults with BD participating as individuals or as parents of at- risk children:

INCLUSION CRITERIA:

* DSM Bipolar Disorder
* Age 18-58
* Be able to complete self-rating forms and to cooperate with other study procedures.
* Medically safe to perform MRI

EXCLUSION CRITERIA:

* Diagnosis of schizophrenia or other current psychosis.
* Claustrophobia or anxiety that prevents participation in MRI
* Any serious medical illness, such as heart, liver, or kidney disease.
* A history of drug or alcohol abuse in the past 90 days.
* Current or past seizure disorder
* Currently unstable hyperthyroidism or hypothyroidism
* Currently receiving medical treatment that would affect mood, such as steroids
* Pregnant or breast-feeding.
* Active suicidal or homicidal thoughts or plans
* NIMH IRP Employee/family member

Healthy volunteer children and adolescents:

INCLUSION CRITERIA:

* Age- and sex- matched to the bipolar patients.
* Have an identified primary care physician.
* Speaks English

EXCLUSION CRITERIA

* I.Q. < 70
* Any serious medical condition or condition that interferes with fMRI scanning
* Pregnancy
* Past or current diagnosis of any anxiety disorder (panic disorder, GAD, Separation Anxiety Disorder, Social Phobia), mood disorder (manic or hypomanic episode, major depression), OCD, PTSD, Conduct Disorder, psychosis, current suicidal ideation, Tourette
* Disorder, Autism Spectrum Disorder or ADHD.
* Substance abuse within two months prior to study participation or present substance abuse
* History of sexual abuse.
* Parent or sibling with Bipolar Disorder, recurrent MDD, or any disorder with psychosis.
* NIMH IRP Employee family member

Parents of healthy volunteer children (Amish and Non-Amish) and Healthy Adults (not parents):

INCLUSION CRITERIA:

* For healthy adults (not parents): Healthy adults age 25-58
* For parents of healthy volunteers: Parents of control subjects as outlined in B above
* Age 25-58
* Speaks English

EXCLUSION CRITERIA:

* IQ< 70
* Any current psychiatric diagnosis
* NIMH IRP Employee/family member

Control subjects with ADHD but not BD:

INCLUSION CRITERIA:

* Age 8-17
* Currently meets DSM-IV criteria for ADHD
* t score >65 on the Connors Parent scales
* Subjects with other psychiatric disorders including anxiety disorders, dysthymic disorder, past major depression, oppositional defiant disorder, tic disorders, and the learning, communication, and elimination disorders may be accepted

EXCLUSION CRITERIA

* IQ<70
* Pregnancy
* Ongoing medical illness or neurological disorder other than ADHD
* Any condition that would interfere with the participants ability to perform fMRI or other research tasks
* Current Major Depression
* Any past or present manic or hypomanic episode.
* NIMH IRP Employee family member

First- and Second-degree relatives of patients with BD:

INCLUSION CRITERIA:

* First degree relatives (parent or sibling) or second-degree relative (grandparent, grandchild, uncle, aunt, nephew, niece, half-sibling) of patients with BD
* Age 3-58

EXCLUSION CRITERIA:

* Active psychosis
* Dementia
* IQ < 70
* Any clinical condition in need of immediate care
* Any chronic medical illness resulting in impaired CNS function
* Any condition that interferes with the participants ability to perform research tasks
* NIMH IRP Employee/family member

Amish Community children with BD:

INCLUSION CRITERIA:

* Age 8-17
* Meet DSM-IV criteria for BD
* Have a primary caregiver who can provide a reliable history
* Be able to complete self-rating forms and to cooperate with other study procedures.

EXCLUSION CRITERIA:

* IQ<70
* Active psychosis
* Any clinical condition in need of immediate care
* Any chronic medical illness resulting in impaired CNS function
* Any condition that would interfere with the participants ability to perform behavioral research tasks
* Limitations with English that would interfere with understanding consent/assent, interview, or task instructions.
* NIMH IRP Employee family member

Amish Community Adults with BD:

INCLUSION CRITERIA:

* DSM-IV Bipolar Disorder
* Age 18-58
* Be able to complete self-rating forms and to cooperate with other study procedures.

EXCLUSION CRITERIA:

* Diagnosis of schizophrenia or other current psychosis.
* Any serious medical illness, such as heart, liver, or kidney disease.
* A history of drug or alcohol abuse in the past 90 days.
* Current or past seizure disorder
* Currently unstable hyperthyroidism or hypothyroidism
* Currently receiving medical treatment that would affect mood, such as steroids
* Active suicidal or homicidal thoughts or plans
* Limitations with English that would interfere with understanding consent/assent, interview, or task instructions.
* NIMH IRP Employee/family member

Amish Community at-risk subjects:

INCLUSION CRITERIA:

* Age 8-17
* Parent or sibling (first-degree relative) diagnosed with BD

EXCLUSION CRITERIA:

* IQ<70
* Active psychosis
* Any clinical condition in need of immediate care
* Any chronic medical illness resulting in impaired CNS function
* Any condition that would interfere with the participants ability to perform behavioral research tasks
* Limitations with English that would interfere with understanding consent/assent, interview, or task instructions.
* NIMH IRP Employee family member

Amish Community healthy volunteer children & adolescents:

INCLUSION CRITERIA:

* Age 8-17
* No serious physical or neurological symptoms or disorder by history

EXCLUSION CRITERIA:

* I.Q. < 70
* Ongoing medical illness
* Neurological disorder (including seizures)
* Past or present substance abuse
* History of sexual abuse
* Limitations with English that would interfere with understanding consent/assent, interview or task instructions
* Past or present psychopathology in control subject or their first-degree relative
* NIMH IRP Employee family member

Amish Community adults who are parents of healthy volunteer children & adolescents, healthy spouses of Amish adults with BD, or parents of adolescents with BD:

INCLUSION CRITERIA:

* Age 18-58
* No serious physical or neurological symptoms or disorder by history
* For Parents of child with BD or spouses of patient with BD: Spouse or offspring with BD

EXCLUSION CRITERIA:

* I.Q. < 70
* Ongoing medical illness
* Neurological disorder (including seizures)
* Past or present substance abuse
* History of sexual abuse
* Limitations with English that would interfere with understanding consent/assent, interview or task instructions
* NIMH IRP Employee/family member
* For Healthy volunteers: Past or present psychopathology in participant or their first-degree relative
* For Parents of healthy volunteer children: Past or present psychopathology as in (4) above.

In addition, children with BD (Section B.1.) who wish to receive treatment, including discontinuation of medication while inpatients on the pediatric behavioral health unit at NIH, may be eligible for treatment if they meet the following additional criteria:

All inclusion criteria for B.1 (above)

Treatment failure as defined by current CGAS score <60

The child s psychiatrist/treating physician agrees that a change in medication regimen is appropriate

EXCLUSION CRITERIA:

All exclusion criteria for B.1 (above)

Any contraindications for MRI scanning, plus claustrophobia or extreme separation anxiety

EXCLUSIONS for MRI Scanning:

* Pregnancy
* Substance abuse within two months of the initial evaluation, since alcohol and abused substances interfere with interpretation of fMRI and cognitive task data.
* Claustrophobia or anxiety that prevents participation in MRI
* Any serious medical condition or condition that interferes with fMRI scanning
* Metal in body which would make having an MRI scan unsafe, such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or if you were a welder or metal worker, since there may be

small metal fragments in the eye

- Unable to lie comfortably on back for up to 90 minutes

Ages: 3 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: There are 11 separate populations being studied in this protocol: 1. Children and adolescents between the ages of 6-17 years old who meet criteria for BSD. 2. Adults between the ages of 18-58 years old who meet criteria for BD, including those age 18-25 with BSD. 3. Control populations of: a) Healthy volunteer children and adolescents between the ages of 3-17 years old, b) Parents of healthy volunteer children or healthy adults in research, c) Children 8-17 years old with attention deficit hyperactivity disorder (ADHD), who do not have a mood disorder. 4. First and second-degree biological relatives of those in (B.1) or (B.2), above, and are between 3-58 years old. 5. A subgroup of these cohorts will be Old Order Amish individuals who fulfill eligibility for (1), (2), (3a), (3b), or (4).
Sampling Method: Non-Probability Sample
Enrollment: 1303 (Actual)
Dates: Start 2000-08-11

PRIMARY OUTCOMES:
Objective 1: clinical manifestations | lifetime of protocol
  (1) clinical interviews [e.g., Schedule for Affective Disorders and Schizophrenia for School-Age Children-present and lifetime version, K-SADS-PL, (Kaufman et al., 1997); Structured Clinical Interview for DSM-IV-TR Axis I Disorders, SCID (First et al., 2002)]; (2) clinical and mood rating assessments (e.g., Children's Depression Rating Scale (Poznanski et al., 1984), Young Mania Rating Scale (Young et al., 1978), Pediatric Anxiety Rating (2002), EMA; (3) episode setting via detailed clinical interview at baseline and every 6 month follow up phone call (4) parent-report and self-report [e.g., The Screen for Child Anxiety Related Emotional Disorders SCARED (Birmaher et al., 1997); Social Responsiveness Scale, SRS (Constantino et al., 2003, Granader et al.); Child Behavior Checklist CBCL (Achenbach, 1991)].
Objective 2: behavioral, neuropsychological, neurophysiological, and neuroanatomical correlates | lifetime of protocol
  1) behavioral performance (e.g., accuracy, response time) on tasks assessing attention, emotion, and attention-emotion interactions; (e.g., Stop/Change task, CPT/Flanker, Decision Making tasks) 2) neuropsychological performance (e.g., performance and verbal IQ) 3) brain activation using functional MRI during tasks assessing attention, emotion, and attention-emotion interactions; 4) structural MRI to examine the size, shape and development of grey matter; 5) Diffusion Tensor Imaging (DTI) to measure white matter track myelination; 6) resting state imaging to test functional connectivity between prefrontal regions and the amygdala
Objective 3: genetic and familial correlates | lifetime of protocol
  (1) clinical interviews [e.g., Schedule for Affective Disorders and Schizophrenia for School-Age Children-present and lifetime version, K-SADS-PL, (Kaufman et al., 1997); Structured Clinical Interview for DSM-IV-TR Axis I Disorders, SCID (First et al., 2002)] to examine the rate of various diagnoses in relatives of individuals with BD (2) genetic material to compare genetic polymorphisms in BSD, their relatives and controls (3) relationship between genetic material and performance on behavioral tasks and activation during fMRI paradigms (4) behavioral performance on standardized paradigms; brain activation using functional MRI; size, shape and development of several ROIs using structural MRI; Diffusion Tensor Imaging (DTI); and, Resting State in individuals with a BD relative

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Leibenluft, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
.We do not plan to make IDP available.

REFERENCES:
- [Background] Geller B, Sun K, Zimerman B, Luby J, Frazier J, Williams M. Complex and rapid-cycling in bipolar children and adolescents: a preliminary study. J Affect Disord. 1995 Aug 18;34(4):259-68. doi: 10.1016/0165-0327(95)00023-g. PMID 8550951
- [Background] Wozniak J, Biederman J, Kiely K, Ablon JS, Faraone SV, Mundy E, Mennin D. Mania-like symptoms suggestive of childhood-onset bipolar disorder in clinically referred children. J Am Acad Child Adolesc Psychiatry. 1995 Jul;34(7):867-76. doi: 10.1097/00004583-199507000-00010. PMID 7649957
- [Background] Faedda GL, Baldessarini RJ, Suppes T, Tondo L, Becker I, Lipschitz DS. Pediatric-onset bipolar disorder: a neglected clinical and public health problem. Harv Rev Psychiatry. 1995 Nov-Dec;3(4):171-95. doi: 10.3109/10673229509017185. PMID 9384947
- [Derived] Chen G, Taylor PA, Reynolds RC, Leibenluft E, Pine DS, Brotman MA, Pagliaccio D, Haller SP. BOLD Response is more than just magnitude: Improving detection sensitivity through capturing hemodynamic profiles. Neuroimage. 2023 Aug 15;277:120224. doi: 10.1016/j.neuroimage.2023.120224. Epub 2023 Jun 15. PMID 37327955
- [Derived] Haller SP, Archer C, Jeong A, Jaffe A, Jones EL, Harrewijn A, Naim R, Linke JO, Stoddard J, Brotman MA. Changes in Internalizing Symptoms During the COVID-19 Pandemic in a Transdiagnostic Sample of Youth: Exploring Mediators and Predictors. Child Psychiatry Hum Dev. 2024 Feb;55(1):206-218. doi: 10.1007/s10578-022-01382-z. Epub 2022 Jul 6. PMID 35794298
- [Derived] Zik J, Deveney CM, Ellingson JM, Haller SP, Kircanski K, Cardinale EM, Brotman MA, Stoddard J. Understanding Irritability in Relation to Anger, Aggression, and Informant in a Pediatric Clinical Population. J Am Acad Child Adolesc Psychiatry. 2022 May;61(5):711-720. doi: 10.1016/j.jaac.2021.08.012. Epub 2021 Aug 23. PMID 34438022
- [Derived] Scheinost D, Dadashkarimi J, Finn ES, Wambach CG, MacGillivray C, Roule AL, Niendam TA, Pine DS, Brotman MA, Leibenluft E, Tseng WL. Functional connectivity during frustration: a preliminary study of predictive modeling of irritability in youth. Neuropsychopharmacology. 2021 Jun;46(7):1300-1306. doi: 10.1038/s41386-020-00954-8. Epub 2021 Jan 21. PMID 33479511
- [Derived] Haller SP, Stoddard J, Pagliaccio D, Bui H, MacGillivray C, Jones M, Brotman MA. Computational Modeling of Attentional Impairments in Disruptive Mood Dysregulation and Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2021 May;60(5):637-645. doi: 10.1016/j.jaac.2020.08.468. Epub 2020 Nov 24. PMID 33242544
- [Derived] Haller SP, Kircanski K, Stringaris A, Clayton M, Bui H, Agorsor C, Cardenas SI, Towbin KE, Pine DS, Leibenluft E, Brotman MA. The Clinician Affective Reactivity Index: Validity and Reliability of a Clinician-Rated Assessment of Irritability. Behav Ther. 2020 Mar;51(2):283-293. doi: 10.1016/j.beth.2019.10.005. Epub 2019 Nov 27. PMID 32138938
- [Derived] Leibenluft E. Chronic irritability in children is not pediatric bipolar disorder: Implications for treatment. Bipolar Disord. 2020 Mar;22(2):195-196. doi: 10.1111/bdi.12881. Epub 2019 Dec 19. No abstract available. PMID 31820531
- [Derived] Linke JO, Adleman NE, Sarlls J, Ross A, Perlstein S, Frank HR, Towbin KE, Pine DS, Leibenluft E, Brotman MA. White Matter Microstructure in Pediatric Bipolar Disorder and Disruptive Mood Dysregulation Disorder. J Am Acad Child Adolesc Psychiatry. 2020 Oct;59(10):1135-1145. doi: 10.1016/j.jaac.2019.05.035. Epub 2019 Jul 19. PMID 31330239
- [Derived] Cardinale EM, Kircanski K, Brooks J, Gold AL, Towbin KE, Pine DS, Leibenluft E, Brotman MA. Parsing neurodevelopmental features of irritability and anxiety: Replication and validation of a latent variable approach. Dev Psychopathol. 2019 Aug;31(3):917-929. doi: 10.1017/S095457941900035X. Epub 2019 May 8. PMID 31064595
- [Derived] Kryza-Lacombe M, Brotman MA, Reynolds RC, Towbin K, Pine DS, Leibenluft E, Wiggins JL. Neural mechanisms of face emotion processing in youths and adults with bipolar disorder. Bipolar Disord. 2019 Jun;21(4):309-320. doi: 10.1111/bdi.12768. Epub 2019 Apr 1. PMID 30851221
- [Derived] Tseng WL, Deveney CM, Stoddard J, Kircanski K, Frackman AE, Yi JY, Hsu D, Moroney E, Machlin L, Donahue L, Roule A, Perhamus G, Reynolds RC, Roberson-Nay R, Hettema JM, Towbin KE, Stringaris A, Pine DS, Brotman MA, Leibenluft E. Brain Mechanisms of Attention Orienting Following Frustration: Associations With Irritability and Age in Youths. Am J Psychiatry. 2019 Jan 1;176(1):67-76. doi: 10.1176/appi.ajp.2018.18040491. Epub 2018 Oct 19. PMID 30336704
- [Derived] Stringaris A, Vidal-Ribas P, Brotman MA, Leibenluft E. Practitioner Review: Definition, recognition, and treatment challenges of irritability in young people. J Child Psychol Psychiatry. 2018 Jul;59(7):721-739. doi: 10.1111/jcpp.12823. Epub 2017 Oct 30. PMID 29083031
- [Derived] Brotman MA, Kircanski K, Leibenluft E. Irritability in Children and Adolescents. Annu Rev Clin Psychol. 2017 May 8;13:317-341. doi: 10.1146/annurev-clinpsy-032816-044941. PMID 28482689
- [Derived] Brotman MA, Kircanski K, Stringaris A, Pine DS, Leibenluft E. Irritability in Youths: A Translational Model. Am J Psychiatry. 2017 Jun 1;174(6):520-532. doi: 10.1176/appi.ajp.2016.16070839. Epub 2017 Jan 20. PMID 28103715
- [Derived] Wiggins JL, Brotman MA, Adleman NE, Kim P, Wambach CG, Reynolds RC, Chen G, Towbin K, Pine DS, Leibenluft E. Neural Markers in Pediatric Bipolar Disorder and Familial Risk for Bipolar Disorder. J Am Acad Child Adolesc Psychiatry. 2017 Jan;56(1):67-78. doi: 10.1016/j.jaac.2016.10.009. Epub 2016 Nov 2. PMID 27993231
- [Derived] Tseng WL, Thomas LA, Harkins E, Stoddard J, Zarate CA Jr, Pine DS, Leibenluft E, Brotman MA. Functional connectivity during masked and unmasked face emotion processing in bipolar disorder. Psychiatry Res Neuroimaging. 2016 Dec 30;258:1-9. doi: 10.1016/j.pscychresns.2016.10.006. Epub 2016 Oct 24. PMID 27814457
- [Derived] Stoddard J, Gotts SJ, Brotman MA, Lever S, Hsu D, Zarate C, Ernst M, Pine DS, Leibenluft E. Aberrant intrinsic functional connectivity within and between corticostriatal and temporal-parietal networks in adults and youth with bipolar disorder. Psychol Med. 2016 May;46(7):1509-22. doi: 10.1017/S0033291716000143. Epub 2016 Feb 29. PMID 26924633
- [Derived] Wiggins JL, Brotman MA, Adleman NE, Kim P, Oakes AH, Reynolds RC, Chen G, Pine DS, Leibenluft E. Neural Correlates of Irritability in Disruptive Mood Dysregulation and Bipolar Disorders. Am J Psychiatry. 2016 Jul 1;173(7):722-30. doi: 10.1176/appi.ajp.2015.15060833. Epub 2016 Feb 19. PMID 26892942
- [Derived] Stoddard J, Sharif-Askary B, Harkins EA, Frank HR, Brotman MA, Penton-Voak IS, Maoz K, Bar-Haim Y, Munafo M, Pine DS, Leibenluft E. An Open Pilot Study of Training Hostile Interpretation Bias to Treat Disruptive Mood Dysregulation Disorder. J Child Adolesc Psychopharmacol. 2016 Feb;26(1):49-57. doi: 10.1089/cap.2015.0100. Epub 2016 Jan 8. PMID 26745832
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-M-0198.html